CLINICAL TRIAL: NCT03816397
Title: Adalimumab in Juvenile Idiopathic Arthritis-associated Uveitis Stopping Trial
Brief Title: Adalimumab in JIA-associated Uveitis Stopping Trial
Acronym: ADJUST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nisha Acharya (Other)
Collaborators: Children's Hospital of Philadelphia (Other); Children's Hospital Medical Center, Cincinnati (Other); Children's Mercy Hospital Kansas City (Other); National Eye Institute (NEI) (NIH); Great Ormond Street Hospital for Children NHS Foundation Trust (Other); University Hospitals Bristol and Weston NHS Foundation Trust (Other); Alder Hey Children's NHS Foundation Trust (Other); Newcastle-upon-Tyne Hospitals NHS Trust (Other); Sheffield Children's NHS Foundation Trust (Other); Cambridge University Hospitals NHS Foundation Trust (Other); Royal Children's Hospital (Other); Norfolk and Norwich University Hospitals NHS Foundation Trust (Other); Vanderbilt University Medical Center (Other); University of California, Davis (Other); University of Texas at Austin (Other); University of Miami (Other); University Hospitals, Leicester (Other); University of Utah (Other); Colorado Retina Associates (Unknown); Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor-Investigator, Nisha Acharya, Director, Uveitis and Ocular Inflammatory Disease Service, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17-23987; UG1EY029658 (NIH)
Record Dates: First submitted 2019-01-22; First posted 2019-01-25 (Actual); Results first posted 2025-03-26 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Uveitis; JIA
Keywords: chronic anterior uveitis; adalimumab; JIA-associated uveitis; stopping
MeSH Terms: conditions — Uveitis; Uveitis, Intermediate | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Continue adalimumab (Active Comparator): Patients randomized to this arm will continue adalimumab at their current weight-based dose administered subcutaneously every other week.
  Interventions: Biological: Adalimumab
- Stop adalimumab (Placebo Comparator): Patients randomized to this arm will receive a volume-matched placebo administered subcutaneously every other week.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Adalimumab — Adalimumab is a fully human monoclonal anti-tumor necrosis factor alpha antibody, a biologic, immunomodulatory drug. Adalimumab 20mg/0.8 mL and 40mg/0.8 mL is a clear, colorless solution provided in a pre-filled syringe for subcutaneous injection. The formulation is adalimumab, mannitol, polysorbate 80, and water for injection Each pre-filled syringe has a fixed 29-gauge thin wall and ½ inch needle with black protective cover and is intended for a single dose to a single patient.
  Other Names: HUMIRA
  Arms: Continue adalimumab
Other: Placebo — The placebo solution is a clear, colorless solution provided in a single-use, pre-filled syringe for subcutaneous injection. The volume-matched (0.8mL) placebo is designed to match the characteristics of the citrate-free adalimumab during injection.
  Arms: Stop adalimumab

SUMMARY:
The proposed study is a stratified, block-randomized, double-masked, controlled trial to determine the feasibility of discontinuing adalimumab treatment in patients with quiescent uveitis associated with juvenile idiopathic arthritis (JIA) or chronic anterior uveitis (CAU).

DETAILED DESCRIPTION:
Background: Juvenile idiopathic arthritis (JIA)-associated uveitis is a chronic pediatric ocular inflammatory condition that can result in visual impairment. Chronic anterior uveitis (CAU) does not have systemic manifestations of disease but presents similarly in the eye and can result in identical visual complications as JIA-associated uveitis. Adalimumab, a tumor necrosis factor (TNF) inhibitor, effectively controls joint and eye inflammation; however, its long-term use may increase the risk of adverse health outcomes and place an undue financial burden on the patient and healthcare system given its high cost. There is great interest for patients to stop adalimumab following remission due to these reasons but there is a lack of information on the ability to maintain control after discontinuing adalimumab.

Methods: The Adalimumab in Juvenile Idiopathic Arthritis-associated Uveitis Trial (ADJUST) is a multi-center international trial that will randomize 118 participants aged 2 years and older with controlled JIA-associated uveitis or chronic anterior uveitis to either continue adalimumab or discontinue adalimumab and receive a placebo. The trial will compare the time to uveitis recurrence between the two groups over 12 months. All participants will receive the standard weight-based dose of adalimumab or placebo: 20 mg biweekly (if < 30 kg) or 40 mg biweekly (if ≥ 30 kg).

Impact: This is the first randomized controlled trial to assess the efficacy of discontinuing adalimumab after demonstrating control of JIA-associated uveitis for at least 12 months. The results of ADJUST will provide information on clinical outcomes to guide clinicians in their decision-making regarding discontinuation of adalimumab.

ELIGIBILITY:
Inclusion Criteria (must meet all of the following to qualify):

* Stated willingness to comply with all study procedures and availability for the duration of the study period
* ≥ 2 years of age
* History of JIA or CAU diagnosed prior to 16 years of age (patient may be older than 16 at time of enrollment)
* Formal diagnosis of JIA-associated uveitis or CAU with no other suspected etiology
* ≥12 consecutive months of controlled ocular inflammation (≤0.5+ anterior chamber cell, ≤0.5+ vitreous haze, no active retinal/choroidal lesions in either eye)
* ≥ 12 consecutive months of controlled arthritis verified by a pediatric rheumatologist, if defined as JIA-associated uveitis
* ≥12 consecutive months of treatment with adalimumab or a biosimilar of adalimumab
* ≥180 days on a stable dose of adalimumab or a biosimilar; must be biweekly dose of either 20mg (if<30kg) or 40mg (if ≥30kg)
* If on a biosimilar of adalimumab, ≥90 days on the biosimilar
* If on concomitant antimetabolite (injectable or oral methotrexate, mycophenolate mofetil, azathioprine, or leflunomide), dose must be ≤25 mg weekly for methotrexate, ≤3 g daily for mycophenolate mofetil, ≤250 mg daily for azathioprine, or ≤20 mg daily for leflunomide; dose and route of administration must be stable for ≥90 days
* If on topical corticosteroids, dose must be ≤2 drops prednisolone acetate 1% or equivalent per day and stable for ≥90 days
* Willingness to limit consumption of alcohol during the study period
* Agreement to avoid live attenuated vaccinations
* Agreement to use highly effective contraception for ≥28 days prior to screening and throughout study period (for males and females of reproductive age)
* Suitable, in the opinion of the Investigator, to continue treatment with adalimumab or placebo per regional labeling
* No contraindications to receive adalimumab as per the local Summary of Product Characteristics (SmPC)

Exclusion Criteria (any one of these excludes the patient):

* Intraocular surgery in the past 90 days or planned surgery in the next 12 months
* Severe cataract or opacity preventing view to the posterior pole in both eyes
* Chronic hypotony (<5 mmHg for ≥90 days) in either eye
* Treatment with oral corticosteroids or intraocular corticosteroid injection within the last 12 months
* Use of NSAID eye drops within the last 90 days
* Acute anterior uveitis characterized by redness and symptoms, including but not limited to floaters, pain, and light sensitivity
* Pregnancy or lactation (a pregnancy test will be conducted at baseline and all follow-up visits for females of reproductive age)
* Presence of intraretinal or subretinal fluid in either eye
* Prior safety or tolerability issues with adalimumab
* History of cancer, active tuberculosis, or hepatitis B
* Other medical condition expected to dictate treatment course during the study
* Any of the following laboratory test results on their most recent tests within the past 90 days prior to screening/enrollment: leukocyte count <2500, platelet count ≤75000, hemoglobin <9.0, Aspartate Aminotransferase (AST) or Alanine Transferase (ALT) ≥ 2 times the upper limit of normal range, creatinine ≥1.5

There are no sex, race, or ethnicity restrictions for this study.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2025-01-23 (Actual); Study Completion 2025-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nisha Acharya, MD MS, Principal Investigator — Principal Investigator
Locations (21):
- United States (11):
  - University of California, Davis, Sacramento, California
  - University of California, San Francisco, San Francisco, California
  - University of Colorado Denver, Aurora, Colorado
  - Colorado Retina Associates, Lakewood, Colorado
  - University of Miami, Miami, Florida
  - Children's Mercy Hospital, Kansas City, Missouri
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas, Austin, Austin, Texas
  - University of Utah Health, Salt Lake City, Utah
- Murdoch Children's Research Institute, Parkville, Victoria, Australia
- United Kingdom (9):
  - University Hospitals Bristol and Weston, Bristol
  - Cambridge University Hospital, Cambridge
  - University Hospitals, Leicester, Leicester
  - Alder Hey Children's Hospital, Liverpool
  - Great Ormond Street Hospital, London
  - Manchester University NHS Foundation Trust, Manchester
  - Great North Children's Hospital, Newcastle upon Tyne
  - Norfolk and Norwich University Hospital, Norwich
  - Sheffield Children's Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jaffe GJ, Dick AD, Brezin AP, Nguyen QD, Thorne JE, Kestelyn P, Barisani-Asenbauer T, Franco P, Heiligenhaus A, Scales D, Chu DS, Camez A, Kwatra NV, Song AP, Kron M, Tari S, Suhler EB. Adalimumab in Patients with Active Noninfectious Uveitis. N Engl J Med. 2016 Sep 8;375(10):932-43. doi: 10.1056/NEJMoa1509852. PMID 27602665
- [Background] Nguyen QD, Merrill PT, Jaffe GJ, Dick AD, Kurup SK, Sheppard J, Schlaen A, Pavesio C, Cimino L, Van Calster J, Camez AA, Kwatra NV, Song AP, Kron M, Tari S, Brezin AP. Adalimumab for prevention of uveitic flare in patients with inactive non-infectious uveitis controlled by corticosteroids (VISUAL II): a multicentre, double-masked, randomised, placebo-controlled phase 3 trial. Lancet. 2016 Sep 17;388(10050):1183-92. doi: 10.1016/S0140-6736(16)31339-3. Epub 2016 Aug 16. PMID 27542302
- [Background] Ramanan AV, Dick AD, Benton D, Compeyrot-Lacassagne S, Dawoud D, Hardwick B, Hickey H, Hughes D, Jones A, Woo P, Edelsten C, Beresford MW; SYCAMORE Trial Management Group. A randomised controlled trial of the clinical effectiveness, safety and cost-effectiveness of adalimumab in combination with methotrexate for the treatment of juvenile idiopathic arthritis associated uveitis (SYCAMORE Trial). Trials. 2014 Jan 9;15:14. doi: 10.1186/1745-6215-15-14. PMID 24405833
- [Background] Vazquez-Cobian LB, Flynn T, Lehman TJ. Adalimumab therapy for childhood uveitis. J Pediatr. 2006 Oct;149(4):572-5. doi: 10.1016/j.jpeds.2006.04.058. PMID 17011337
- [Background] Chang CY, Meyer RM, Reiff AO. Impact of medication withdrawal method on flare-free survival in patients with juvenile idiopathic arthritis on combination therapy. Arthritis Care Res (Hoboken). 2015 May;67(5):658-66. doi: 10.1002/acr.22477. PMID 25220674
- [Background] Baszis K, Garbutt J, Toib D, Mao J, King A, White A, French A. Clinical outcomes after withdrawal of anti-tumor necrosis factor alpha therapy in patients with juvenile idiopathic arthritis: a twelve-year experience. Arthritis Rheum. 2011 Oct;63(10):3163-8. doi: 10.1002/art.30502. PMID 21702011
- [Background] Shakoor A, Esterberg E, Acharya NR. Recurrence of uveitis after discontinuation of infliximab. Ocul Immunol Inflamm. 2014 Apr;22(2):96-101. doi: 10.3109/09273948.2013.812222. Epub 2013 Jul 22. PMID 23876234
- [Background] Acharya NR, Ebert CD, Kelly NK, Porco TC, Ramanan AV, Arnold BF; ADJUST Research Group. Discontinuing adalimumab in patients with controlled juvenile idiopathic arthritis-associated uveitis (ADJUST-Adalimumab in Juvenile Idiopathic Arthritis-associated Uveitis Stopping Trial): study protocol for a randomised controlled trial. Trials. 2020 Oct 27;21(1):887. doi: 10.1186/s13063-020-04796-z. PMID 33109240
- [Result] Acharya NR, Ramanan AV, Coyne AB, Dudum KL, Rubio EM, Woods SM, Guly CM, Moraitis E, Petrushkin HJD, Armon K, Puvanachandra N, Choi JT, Hawley DP, Arnold BF; ADJUST Study Group. Stopping of adalimumab in juvenile idiopathic arthritis-associated uveitis (ADJUST): a multicentre, double-masked, randomised controlled trial. Lancet. 2025 Jan 25;405(10475):303-313. doi: 10.1016/S0140-6736(24)02468-1. PMID 39863370

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled from March 3, 2020, to Feb 14, 2024, at 20 ophthalmology and rheumatology clinical sites across the United States, the United Kingdom, and Australia.
Groups:
- Continue Adalimumab: Patients randomized to this arm will continue adalimumab at their current dose administered subcutaneously every other week.
- Stop Adalimumab: Patients randomized to this arm will receive a volume-matched placebo (0.8mL) administered subcutaneously every other week.
Period: Overall Study
Arm/Group | Continue Adalimumab | Stop Adalimumab
Started | 43 | 44
Completed | 29 | 37
Not Completed | 14 | 7
Not completed — Censored at interim analysis date. | 13 | 6
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Stop Adalimumab: Patients randomized to this arm will receive a volume-matched placebo (0.8 mL) administered subcutaneously every other week.
- Total: Total of all reporting groups
Arm/Group | Continue Adalimumab | Stop Adalimumab | Total
Number analyzed (Participants) | 43 | 44 | 87
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 12.56 [9.44 to 15.81] | 12.26 [9.39 to 13.42] | 12.31 [9.39 to 15.28]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 32 | 64
  Male | 11 | 12 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 8 | 14
  Not Hispanic or Latino | 35 | 28 | 63
  Unknown or Not Reported | 2 | 8 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 34 | 33 | 67
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 1 | 4 | 5
Region of Enrollment [Number; unit: participants]
  United States | 14 | 14 | 28
  United Kingdom | 27 | 27 | 54
  Australia | 2 | 3 | 5
Conventional DMARD Use [Count of Participants; unit: Participants]
  Azathioprine | 1 | 3 | 4
  Leflunomide | 2 | 1 | 3
  Methotrexate (oral) | 13 | 9 | 22
  Methotrexate (subcutaneous) | 14 | 15 | 29
  Mycophenolate mofetil | 1 | 3 | 4
  None | 12 | 13 | 25
Arthritis category [Count of Participants; unit: Participants]
  None; chronic anterior uveitis | 7 | 7 | 14
  Oligoarthritis | 29 | 29 | 58
  Polyarthritis | 7 | 6 | 13
  Psoriatic arthritis | 0 | 1 | 1
  Undifferentiated arthritis | 0 | 1 | 1
Age at diagnosis of juvenile idiopathic arthritis, years [Median (Inter-Quartile Range); unit: years] | 2.77 [2.30 to 4.52] | 3.71 [2.36 to 6.18] | 3.30 [2.32 to 5.59]

OUTCOME MEASURES:

1. Primary Outcome: Time to Treatment Failure
Description: Treatment failure is defined by recurrence of ocular inflammation in at least one eye as follows:
  * 3+ anterior chamber (AC) for a single visit
    •>0.5+ anterior chamber (AC) cell for ≥28 days
  * 2-step increase in AC cell observed at two separate visits ≥7 days apart
    * 0.5+ vitreous haze, active retinal or choroidal inflammation, or macular edema observed at a single visit. Treatment failure can also be declared by recurrence of joint inflammation that is persistent and severe enough to necessitate unmasking to manage the arthritis recurrence.
  Time (days) from all participants is included in the analysis.
Time Frame: From baseline until 48 weeks post-randomization
Population: Two patients dropped out of the trial before reaching the primary endpoint (one in each group). The length of time that these patients participated in the trial before dropout is included in the primary outcome analysis given the nature of survival analyses. Patients still in active follow-up who had not yet reached the primary endpoint (13 in the adalimumab group and six in the placebo group) were censored at the interim analysis date, Feb 14, 2024. No patients were lost to follow-up.
Measure: Median (Inter-Quartile Range); unit: Time to treatment failure (days)
Arm/Group | Continue Adalimumab | Stop Adalimumab
Number analyzed (Participants) | 43 | 44
Time to treatment failure (days) | NA [NA to NA] — Data are not available because a median time to treatment failure and Inter-Quartile Range (IQR) could not be calculated due to an insufficient number of participants with events. | 119 [84 to 243]
Statistical Analysis 1: Comparison: Continue Adalimumab vs Stop Adalimumab; A Cox proportional hazards regression was used to compare time to treatment failure between the adalimumab and placebo groups up to the primary endpoint of 48 weeks, with country and conventional DMARD use included as fixed effects in the model. The null hypothesis was an hazard ratio (HR) of 1. Hypothesis testing was based on a permutation test of the log hazard ratio (100,000 replicates). The model was checked for the assumption of proportional hazards by assessing Schoenfeld residuals; Test type: Superiority — A sample size of 118 subjects (59 in each group) provides 88% power to detect a hazard ratio of 2.0 for the time to treatment failure comparing the group randomized to discontinue adalimumab to the group randomized to continue using adalimumab, assuming a median time until treatment failure of 10 weeks in the group that discontinues adalimumab (Arm 1) and of 20 weeks in the group that continues on adalimumab (Arm 2), an equal allocation between groups, and a 10% total loss to follow-up; p < 0.0001, Log Rank — A priori threshold for statistical significance was <0.05; Hazard Ratio (HR) = 8.7, 95% CI 2-sided [3.6 to 21.2] — For the HR, the numerator is the placebo group (stop adalimumab) and the denominator is the adalimumab group (continue adalimumab)

ADVERSE EVENTS:
Time Frame: Adverse events shown were reported before or at the primary endpoint (treatment failure or censoring at 48 weeks).
Groups:
- Continue Adalimumab: Patients randomized to this arm will continue adalimumab at their current weight-based dose, administered subcutaneously every other week.
Arm/Group | Continue Adalimumab | Stop Adalimumab
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/44
Serious Adverse Events (participants affected / at risk) | 4/43 | 0/44
Other Adverse Events (participants affected / at risk) | 34/43 | 29/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Continue Adalimumab (N=43) | Stop Adalimumab (N=44)
Surgery for torted cyst of Morgagni (Surgical and medical procedures) | 1 (1) | 0 (0)
Shortness of breath at rest; suspected to be anxiety-related (Psychiatric disorders) | 1 (1) | 0 (0)
Over 5 times the upper limit of normal for alanine aminotransferase (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Planned orthognathic surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Continue Adalimumab (N=43) | Stop Adalimumab (N=44)
Allergic reaction (Respiratory, thoracic and mediastinal disorders) | 5 (10) | 1 (1)
COVID-19 (Infections and infestations) | 12 (15) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (8) | 3 (4)
Ear infection (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 15 (28) | 8 (12)
Fever (Infections and infestations) | 8 (8) | 2 (2)
Influenza (Infections and infestations) | 3 (3) | 1 (1)
Headache (General disorders) | 17 (24) | 10 (20)
Gastrointestinal related (Gastrointestinal disorders) | 24 (51) | 17 (19)
Mood changes (Psychiatric disorders) | 6 (7) | 3 (4)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (2)
Impaired neurological function (Nervous system disorders) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Sinus infection (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Skin infection (Infections and infestations) | 4 (5) | 3 (4)
Upper respiratory infection (Infections and infestations) | 9 (16) | 7 (8)
Other infection‡‡ (Infections and infestations) | 4 (5) | 4 (5)
Atypical haemoglobin (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atypical leukocyte count (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Atypical aspartate aminotransferase or alanine aminotransferase (Blood and lymphatic system disorders) | 2 (3) | 0 (0)
Ocular hypertension (Eye disorders) | 1 (1) | 2 (4)
Other ocular event (Eye disorders) | 4 (4) | 4 (4)
Other events (General disorders) | 14 (31) | 9 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-02-14): https://cdn.clinicaltrials.gov/large-docs/97/NCT03816397/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-14): https://cdn.clinicaltrials.gov/large-docs/97/NCT03816397/SAP_001.pdf